CLINICAL TRIAL: NCT00617214
Title: Evaluation of Treatment Outcomes in Schizophrenic Patients Taking Part in the Integrated Care Program - a Single-country, Multi-centre Non-interventional Study
Brief Title: Schizophrenic Patients Taking Part in Integrated Care Program
Acronym: CARE I
Status: Terminated | Type: Observational
Why Stopped: Difficulty finding eligible sites/patients:current situation in health policy cause negative effects on existing/planned contracts for integrated care programs
Sponsor: AstraZeneca (Industry)
Collaborators: acromion GmbH (Industry)
Other Study IDs: NIS-NDE-SER-2007/1
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2008-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreni-form Disorder; Delusional Disorder; Psychotic Disorder Not Otherwise Specified
Keywords: Schizophrenia; Integrated care program; Seroquel
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All: Schizophrenic outpatients who are treated with Seroquel IR and who are additionally intended to start with an integrated care program

SUMMARY:
Purpose of this non-interventional study (NIS) is to assess the effect of the participation in an integrated care program on treatment outcomes in patients treated with Seroquel for schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients suffering from schizophrenia, schizoaffective disorder, schizophreni-form disorder, delusional disorder or psychotic disorder not otherwise specified
* Age 18 - 65 years
* Current stable treatment with Seroquel according to SmPC since at least 2 months
* Given consent to take part in an integrated care program prior to study startWritten informed consent to take part in this NIS

Exclusion Criteria:

* Presence of any contraindication as described in the SmPC
* Cancellation of participation in the integrated care program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient department from clinics or private practices
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Subjective Well-Being measured via SWN patient questionnaire | 6 month period of observation,4 assessments

SECONDARY OUTCOMES:
Quality of Life and patient's satisfaction measured by Q-LES-Q-18 and CSQ-8 | 6 month period of observation, 1 assessment at end of NIS
Symptomatic and functional outcome measured by CGI-S, PANSS-8, GAF, EQ-5D and VOI | 6 month period of observation, 4 assesments
Compliance and health economic aspects measured by MARS, days of hospitalization, productivity loss | 6 month period of observation, 4 assesments

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Liedtke, MD, Study Director — AstraZeneca; Martin Lambert, PD, MD, Principal Investigator — University of Hamberg
Locations (14):
- Germany (14):
  - Research Site, Ahrweiler
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Hamburg
  - Research Site, Mannheim
  - Research Site, Mittweida
  - Research Site, München
  - Research Site, Münster
  - Research Site, Oldenburg
  - Research Site, Ottobrunn bei München
  - Research Site, Spremberg
  - Research Site, Stolberg
  - Research Site, Werneck
  - Research Site, Zittau